CLINICAL TRIAL: NCT06098482
Title: A Prospective, Repeated-measures Investigation to Validate Digital Speech Perception Endpoints in Adult Cochlear Implant Recipients Using the Mobile Research App: a Master Umbrella Investigation
Brief Title: An Investigation to Validate Speech Perception Assessment for Adult Cochlear Recipients Using a Mobile Research App
Acronym: VALDE-MU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: AI5841
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Delivery of speech perception materials in-clinic using the Mobile Research App (MRA) (Experimental): Cochlear implant recipients will participate in this arm (sub-investigation AI5841A).
  Interventions: Device: Mobile Research App (MRA); Other: SOC/validated delivery of the speech perception test material
- Delivery of speech perception materials in-clinic and at home using the Mobile Research App (MRA) (Experimental): Cochlear implant and hearing aid recipients will participate in this arm (sub-investigation AI5841B).
  Interventions: Device: Mobile Research App (MRA); Other: SOC/validated delivery of the speech perception test material

INTERVENTIONS:
Device: Mobile Research App (MRA) — The MRA (research tool) is a platform used for the delivery of speech perception material in-clinic outside the sound booth or in the home of the hearing-impaired recipients. The MRA speech testing module delivers speech material via streaming to the single implanted ears of cochlear implant recipients. The recipient listens to the speech material and responds with what was heard via the app. Speech is streamed via Bluetooth from the iOS device to the sound processor of the CI-recipient.
Other: SOC/validated delivery of the speech perception test material — This involves the delivery of speech perception test material in the sound booth in a clinic.

SUMMARY:
The study is a feasibility, prospective, repeated-measures, multi-country, multi-centre, study of the Mobile Research App to measure and validate speech perception endpoints in adult cochlear implant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older.
* Uses a hearing device or devices (hearing aid/s and/or cochlear implant/s).
* Fluent speaker in the language used to assess clinical performance as judged by the investigator.
* Willing and able to provide written informed consent.

Exclusion Criteria:

* Unable or unwilling to comply with the requirements of the clinical investigation as determined by the Investigator.
* Investigator site personnel directly affiliated with this study and/or their immediate families; immediate family is defined as a spouse, parent, child, or sibling.
* Cochlear employees or employees of Contract Research Organisations or contractors engaged by Cochlear for the purposes of this investigation.
* Currently participating, or participated within the last 30 days, in another interventional clinical investigation/trial involving an investigational drug or device (unless the other investigation was/is a Cochlear sponsored investigation and determined by the investigator or Sponsor to not impact this investigation).
* Women who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2024-02-05 (Actual); Primary Completion 2027-05-02 (Estimated); Study Completion 2027-05-02 (Estimated)

PRIMARY OUTCOMES:
Percent correct performance for the test and retest runs of speech perception ability | 1 day - immediately post screening.
  To determine if test-retest reliability with a correlation greater than or equal to 0.8 can be achieved for speech perception ability measured on the MRA outside the sound booth, percent correct performance for the test and retest runs of the speech perception ability will be compared.
  Scoring: Percentage correct
  Range: 0-100%, higher scores equal better performance

CONTACTS AND LOCATIONS:
Locations (4):
- Denver Research and Technology Labs, Lone Tree, Colorado, United States
- HEARnet Clinical Studies, Melbourne, Victoria, Australia
- Belgium (2):
  - European Institute for Otorhinolaryngology (EIORL) ENT department Sint-Augustinus Antwerp, Antwerp, Antwerp
  - Hoorzorg van Looveren, Wommelgem, Antwerp

IPD SHARING:
Plan to Share IPD: No